CLINICAL TRIAL: NCT06430125
Title: Clinical Study Evaluating the Nephroprotective Effect of Nicorandil in Patients With Type 2 Diabetes Mellitus
Brief Title: Nephroprotective Effect of Nicorandil in Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Atta Ali El-Hazzab, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nicorandil Nephroprotective
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — Nicorandil; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): this group will include 23 patients who will receive metformin 2gm/day. The initial dose of metformin will be 1 g/day taken orally with the meal. After 7 days (week 1), the dose will be up titrated to daily dose of 2,000 mg/day. Treatment duration will be 12 weeks .
- Nicorandil group (Active Comparator): this group will include 23 patients who will receive a combination of metformin 2g/day and nicorandil 10 mg twice daily. The initial dose of metformin will be 1 g/day taken orally with the meal. After 7 days (week 1), the dose will be uptitrated to daily dose of 2,000 mg/day. Treatment duration will be 12 weeks .
  Interventions: Drug: Nicorandil 10 MG Oral Tablet

INTERVENTIONS:
Drug: Nicorandil 10 MG Oral Tablet — Nicorandil 10 MG oral tablet twice daily
  Arms: Nicorandil group

SUMMARY:
This study aims to evaluate the possible nephroprotective effect of nicorandil in patients with type 2 diabetes mellitus .

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with T2DM with diet control and good glycemic index ( Hb A1C< 7 )
* Age range between 18 and 60 years old.
* Both sexes.
* Stage 1and Stage 2 CKD according to KDIGO .
* Controlled HTN .

Exclusion Criteria:

* Pregnant and lactating females.
* Patients with hypersensitivity to nicorandil.
* Other Causes of CKD or Nephropathy eg : Uncontrolled HTN , Renal Malignancy , collagen disease as Amyloidosis and some autoimmune disease as ( SLE and Rh.fever ) .
* Uncontrolled HTN and its antihypertensive medications ( ACEI , ARB ) and other antihypertensive medications .
* Patients receiving nephrotoxic drugs as aminoglycosides, non-steroidal anti inflammatory drugs and contrast media.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
prevention of progression of kidney disease as measured by KDIGO. | 12 weeks
  Patients wii undergo clinical assesment for progression of diabetic nephropathy as measured by KDIGO at baseline and after 12 weeks

SECONDARY OUTCOMES:
change in the serum concentrations of Kidney injury molecule 1(Kim-1). | 12 weeks
  Venous blood will be collected before treatment and after 12 week .
change in the serum concentrations of Interleukin 18 (IL-18). | 12 weeks
  Venous blood will be collected before treatment and after 12 week .
change in the serum concentrations of Nitric oxide (NO). | 12 weeks
  Venous blood will be collected before treatment and after 12 week .

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, EL Gharbia, Egypt